CLINICAL TRIAL: NCT05177601
Title: A Randomized Sham and Placebo-controlled Trial of Adjunctive D-cycloserine in Repetitive Transcranial Magnetic Stimulation for Obsessive Compulsive Disorder
Brief Title: iTBS-DCS in Obsessive Compulsive Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB21-0265
Record Dates: First submitted 2021-03-22; First posted 2022-01-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- TMS+DCS (Active Comparator): The Transcranial Magnetic Stimulation (TMS) involves magnetic stimulation of the brain to the left medial prefrontal cortex (mPFC) daily for four weeks. The stimulation is intermittent Theta-Burst (iTBS).
  Participants will orally ingest a capsule containing 100mg of the antibiotic d-cycloserine (DCS) daily (Monday-Friday) for 4 weeks of rTMS treatment (20 sessions) one hour prior to rTMS treatment.
  Interventions: Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS); Drug: D-cycloserine
- TMS+Placebo (Active Comparator): The Transcranial Magnetic Stimulation (TMS) involves magnetic stimulation of the brain to the left medial prefrontal cortex (mPFC) daily for four weeks. The stimulation is intermittent Theta-Burst (iTBS).
  Participants will orally ingest a capsule identical to that containing the study medication, however this capsule will contain a placebo. They will ingest this capsule daily (Monday-Friday) for 4 weeks of rTMS treatment (20 sessions) one hour prior to rTMS treatment.
  Interventions: Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS); Drug: Placebo oral capsule
- shamTMS+DCS (Sham Comparator): Sham rTMS treatment involves scalp stimulation with no magnetic pulse daily for four weeks (20 sessions). Sham rTMS involves only the click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered to the brain.
  Participants will orally ingest a capsule containing 100mg of the antibiotic d-cycloserine (DCS) daily (Monday-Friday) for 4 weeks of rTMS treatment (20 sessions) one hour prior to rTMS treatment.
  Interventions: Device: Sham rTMS; Drug: D-cycloserine
- shamTMS+placebo (Placebo Comparator): Sham rTMS treatment involves scalp stimulation with no magnetic pulse daily for four weeks (20 sessions). Sham rTMS involves only the click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered to the brain.
  Participants will orally ingest a capsule identical to that containing the study medication, however this capsule will contain a placebo. They will ingest this capsule daily (Monday-Friday) for 4 weeks of rTMS treatment (20 sessions) one hour prior to rTMS treatment.
  Interventions: Device: Sham rTMS; Drug: Placebo oral capsule

INTERVENTIONS:
Device: iTBS repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a non-invasive procedure in which cerebral electrical activity is influenced by a rapidly changing magnetic field. The magnetic field is created by a plastic-encased coil which is placed over the patient's scalp. The magnetic field can be directed onto specific areas of the brain. rTMS can modulate cerebral activity by low or high frequencies. Over time, the magnetic field pulses can gradually change the activity level of the stimulated brain region and help symptoms of mood disorders.
  Other Names: MAGPRO X100 stimulator
  Arms: TMS+DCS; TMS+Placebo
Device: Sham rTMS — Sham rTMS involves a click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered.
  Other Names: MAGPRO X100 stimulator
  Arms: shamTMS+DCS; shamTMS+placebo
Drug: D-cycloserine — Daily oral D-cycloserine 100mg during TMS treatments (20 days).
  Other Names: Seromycin
  Arms: TMS+DCS; shamTMS+DCS
Drug: Placebo oral capsule — Daily oral placebo during the TMS treatments (20 days).
  Arms: TMS+Placebo; shamTMS+placebo

SUMMARY:
Obsessive Compulsive Disorder (OCD)is a common and debilitating illness. For an unacceptable proportion of patients, depressive symptoms remain impairing despite multiple treatments.

In August 2018, the FDA approved transcranial magnetic stimulation (TMS) for the treatment of OCD based on a large study demonstrating efficacy. Our neurophysiological data and clinical data in depression suggests that we can enhance the effects of TMS by using an adjunctive medication called D-Cyloserine (DCS, 100mg) in conjunction with stimulation. The mechanism by which this is achieved is called synaptic plasticity, or the activity dependent changes that occur with brain stimulation.

Research Question and Objectives: To conduct a randomized sham- and placebo-controlled trial of DCS in adjunct with rTMS in OCD. Participants will be randomized to receive 100mg of DCS or placebo together with TMS.

DETAILED DESCRIPTION:
Methods: Eighty one patients (males and females aged 18-65, with a score ≥20 on the Yale-Brown Obsessive Compulsive Scale, stable selective serotonin reuptake inhibitors or cognitive behavioral therapy for 2 months) will be recruited. Patients will be randomized 2:2:1:1 TMS+DCS, TMS+Placebo, Sham+DCS or Sham+Placebo. Participants who do not have recent bloodwork will have laboratory tests to rule out haematological, hepatic, and renal disease, and participants will be screened for suicidal ideation. The dose of DCS will be 100mg, taken daily for four weeks. Clinical outcomes will be quantified using the Yale-Brown Obsessive Compulsive Scale, a gold standard clinician rated instrument for OCD, as well as measures of depression and anxiety. Participants will complete a short battery of cognitive tests and questionnaires to measure self-reported symptoms of depression, anxiety and quality of life. Fecal samples will be taken at baseline, week 4 and week 8 to characterize any changes in the microbiome. Participants clinical symptoms will be evaluated again one-month after treatment. At this time, all participants who received sham-rTMS will be offered an additional 4 weeks of open label rTMS.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 65 years
2. are competent to consent to treatment
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of DSM-5 criteria Obsessive Compulsive Disorder.
4. have failed to achieve a clinical response to one adequate trial of serotonin reuptake inhibitor or cognitive behavioral therapy with an adequate trial of 2 months medication within the current episode, or been unable to tolerate antidepressant medications.
5. have a score ≥ 20 on the YBOCS.
6. have had no change in dose, or initiation of any psychotropic medication in the 8 weeks prior to randomization
7. are able to adhere to the treatment schedule
8. pass the TMS adult safety screening (TASS) questionnaire

Exclusion Criteria:

1. Allergy to cycloserine.
2. have an alcohol or substance use disorder within the last 3 months
3. have suicidal ideation (score of 4 ≥ on item 10 of MADRS)
4. are at a significant risk of harm to themselves or others
5. Current symptoms of psychosis
6. History of psychosis
7. are currently pregnant , breast feeding or plan to become pregnant
8. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of other primary psychiatric diagnoses as assessed by a study investigator to be primary and causing greater impairment than Major Depressive Disorder.
9. have failed a course of ECT in the current episode. Previous ECT treatment outside of the current episode does not influence inclusion.
10. history of non-response to rTMS treatment.
11. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of epilepsy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
12. have concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
13. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
14. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
15. are currently (or in the last 4 weeks) taking lorazepam or any other benzodiazepine due to the potential to limit rTMS efficacy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (YBOCs) | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Change in severity of Obsessive Compulsive Disorder (OCD) symptoms as measured by the YBOCS, a clinician-rated instrument. Scores on the YBOCS range from 0 (no Symptoms) to 40 (Extreme Symptoms). Ranges of severity are: 0-7 Subclinical range, 8-15 Mild, 16-23 Moderate, 24-31 Severe, and 32-40 Extreme.

SECONDARY OUTCOMES:
Clinical Remission | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  score ≤12 on the YBOCs
Clinical Response | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  ≥30% reduction in YBOCS scores from baseline
Montgomery-Asberg Depression Rating Scale (MADRS) | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Change in severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Change in self reported anxiety symptoms | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Anxiety symptoms will be assessed using the 7 item Generalized Anxiety Disorder (GAD-7) questionnaire. The GAD-7 measures self-reported feelings of anxiety within the last 2 weeks. Scores range from 0-21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
Change in quality of Life as measured by the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The WHOQOL-BREF is a self-reported questionnaire which assesses individual's perception of their quality of life across 4 domains; physical health, psychological, social relationships and environment. Domains scores are calculated to range from 0-20 and scaled in a positive direction (ie. higher scores denote higher quality of life).
Change in self reported depressive symptoms as measured by The Quick Inventory of Depressive Symptomatology (QIDS) | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The Quick Inventory of Depressive Symptomatology (QIDS) rates depression symptoms via self-assessment.Severity of depression can be judged based on the total score.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
Change in self reported measures of workplace productivity | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Productivity will be assessed using the Lam Employment Absence and Disability Scale (LEAPS). The LEAPS is a 10-item, self-rated scale and provides information on how participants are functioning at work. Scores range from 0 - 28, with higher scores representing more severe work impairment.
Clinical Global Impression- Severity | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The CGI-Severity scale is clinician rated from 1-7 representing 'Not at all ill' to 'Severely ill'.
Clinical Global Impression- Improvement | Administered at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The CGI-Improvement scale is a clinician rated 1-7, representing the range between 'Very much improved' and 'Very much worse' from the baseline visit.
Stool samples- microbiome analysis | Samples will be collected at baseline, after TMS treatment (week 4) and 4 weeks after completion of TMS (week 8)
  Microbiome analysis will include α-diversity metrics for each sample and β-diversity measures (weighted and unweighted unifrac, Bray-Curtis, nonmetric multidimensional scaling) and other statistical analysis using QIIME and PhyloSeq. Association of specific taxa and co-occurrence of taxa with sample groups will be examined with ANOVA, the G test of independence, or a paired t-test in QIIME. Sequence data will be assembled and analyzed with the QIIME package. Statistical significance of depression-associated signature profiles will be identified by multivariate statistics (PC-ORD software, R statistical package). Microbial 16S rRNA gene sequence libraries will be compared for distinct microbial patterns.
Stool samples- metabolomics | Samples will be collected at baseline, after TMS treatment (week 4) and 4 weeks after completion of TMS (week 8)
  Changes in fecal metabolomics will be assessed. Fecal supernatants will be removed and filtered through 0.2 μm membrane filters. The fecal sample will be transferred to a standard NMR tube for 1H-NMR spectral analysis on a 500 MHz Inova spectrometer. Spectral fitting for metabolites will be done using the standard Chenomx 500 MHz metabolite library. Typically, 90% of visible peaks are assigned to a compound and more than 90% of the spectral area can be routinely fit using the Chenomx spectral analysis software.
Change in Cognitive Function - THINC-it- PDQ-5 | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The cognitive questionnaire is called the Perceived Deficits Questionnaire - 5 item scale (PDQ-5). The questionnaire assesses self perceived cognition by asking questions about attention/concentration, retrospective memory, prospective memory, and planning/organization.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Choice Reaction Time | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The first objective cognitive test is called "spotter" and measures choice reaction time by calculating the total time that elapses between the presentation of a stimulus and the occurrence of a response in a task that requires a participant to make one of two different responses depending on which stimuli is presented.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Working Memory | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The second objective cognitive test is called "Symbol Check" and is an n-back test. N-back tests measure working memory by presenting the subject with a sequence of stimuli, and the task consists of selecting the stimuli that was presented n steps earlier in the sequence.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Digit Symbol Substitution | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The third objective cognitive test is called "CodeBreaker" and is a Digit Symbol Substitution Test (DSST). DSST involves a key consisting of the numbers 1-6, each paired with a unique symbol. Below the key are a series of the numbers 1-6 in random order and repeated several times. Subjects must select the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Trail Making Test part B | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The fourth objective cognitive test is called "Trails" and is a version of the Trail Making Test part B (TMT-B). The subject is presented with numbers and letters in circles placed in random array on the screen. The subject must draw a line from one circle to the next in ascending order; however, s/he must alternate the circles with numbers in them and circles with letters in them (ie, 1-A-2-B-3-C etc). The TMT is a timed test and the goal is to complete the tests accurately and as quickly as possible.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Implicit Suicidality | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Death Implicit Association Test (D-IAT) is a behavioral test that measures the strength of automatic (implicit) associations between concepts in people's minds relying on latency measures in a simple sorting task. The strength of an association between concepts of "death" and "ones self" is measured by the standardized mean difference score of the 'hypothesis-inconsistent' pairings and 'hypothesis-consistent' pairings
Wisconsin Card Sorting Task (WCST) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The WCST is a neuropsychological instrument used to measure the executive functions, reportedly sensitive to brain dysfunction affecting the frontal lobes.
Stop Signal Task | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  The stop-signal reaction time in the Stop-Signal Task. The stop signal reaction time ranges from 50 to 250, where greater values represent worse outcome (i.e, increased motor impulsivity).
Change in self reported cognitive failures as measured by The Cognitive Failures Questionnaire (CFQ) | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The Cognitive Failures Questionnaire (CFQ) is used to assess the frequency with which people experienced cognitive failures, such as absent-mindedness, in everyday life -- slips and errors of perception, memory, and motor functioning.
  Individuals are asked to rate how often in the past 6 months they have experienced different cognitive failures from "never "(0) to "very often" (4). The sum of the ratings of the 25 individual items yields a score from 0-100, with higher scores indicating more cognitive failures.
VAS for General Health | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  A Visual Analog Scale (VAS) will ask participants how good or bad their health is today. This scale is numbered from 0 to 100. 100 indicates the best health they can imagine. 0 indicates the worst health they can imagine.
Change in suicidal intentions | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The Scale for Suicide Ideation (SSI) is a brief 19-item scale that assesses the person's current intensity of attitudes, plans, and behaviors to commit suicide. Each question has 3 answer choices. The answer choice suggesting the least suicide intentions is scored as 0, and answer choice suggesting the most suicide intentions are scored as 2.
  Total score is determined based on the sum of all individual scores.
Change in severity of skin-picking symptoms | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The Yale-Brown Obsessive Compulsive Scale Modified for Neurotic Excoriation (NE-YBOCS) is a 10-item instrument used to assess severity of skin picking disorder symptoms during the preceding seven days. Responses to the 10 items are coded on a 4-point scale and summed to produce a composite score ranging from 0 to 40, with higher scores reflecting greater illness severity.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Daily Monday-Friday throughout study (4 weeks)
  Adverse events will be tracked and recorded
Side Effects | The TSES will be administered at baseline, and weekly throughout study (Week 1, Week 2, Week 3, Week 4), and at follow up (week 8)
  Side effects will be tracked through the Toronto Side Effects Scale (TSES). The TSES is a self reported questionnaire that assesses incidence, frequency, and severity of central nervous system, gastrointestinal, and sexual side effects. Individuals will be asked to rate frequency of each symptom within the last week on a 5-point scale, from "Never" (1) to "Everyday" (5). Severity of each symptom is similarly rated on a 5-point scale, from "No trouble" (1) to "Extreme Trouble" (5).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No